CLINICAL TRIAL: NCT03694132
Title: Evaluation and Characterization of Infraclinical Sensory Deficits in Amyotrophic Lateral Sclerosis by Brain Imaging and Electrophysiology
Brief Title: Brain Excitability and Connectivity in Sensory-motor Pathways in ALS
Acronym: SOM_ALS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: C17-70
Record Dates: First submitted 2018-09-28; First posted 2018-10-03 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2021-09

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Brain excitability; Brain connectivity; Motor cortex; Somatosensory cortex
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Intervention Model Description: patients vs. health subjects
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- functional MRI (Experimental): a group of patients with ALS and a group of gender and age matched healthy subjects will have functional MRI acquisition conditioned by electrical and mechanical stimuli of ADM proprioceptors
  Interventions: Device: functional MRI
- structural MRI (Experimental): a group of patients with ALS and a group of gender and age matched healthy subjects will have diffusion MRI acquisition to evaluate their brain structures
  Interventions: Device: structural MRI
- EEG/MEG (Experimental): a group of patients with ALS and a group of gender and age matched healthy subjects will have functional MRI acquisition conditioned by electrical stimuli of ADM proprioceptors
  Interventions: Device: EEG/MEG

INTERVENTIONS:
Device: functional MRI — conditioning brain activity with peripheral stimulations
  Arms: functional MRI
Device: structural MRI — diffusion MRI and tractography for evaluating the brain structures
  Arms: structural MRI
Device: EEG/MEG — conditioning brain activity with peripheral stimulations
  Arms: EEG/MEG

SUMMARY:
The main objective is to determine the origin of somatosensory alteration in patients with ALS and to evaluate its impact on brain activity by coupling different imaging modalities and indirect electrophysiology.

The secondary objective is to evaluate whether the observed functional changes in MEG / EEG and functional MRI correlate with structural lesions revealed with diffusion MRI (anatomo-functional connectivity of the brain).

DETAILED DESCRIPTION:
Somatosensory evoked potentials (SEPs) produced by ulnar nerve electrical stimulation will be collected with combined MEG and EGG.

Functional MRI will be performed during electrical stimulation of ulnar nerve and during mechanical vibration of ADM tendon.

Brain diffusion MRI will be performed. Anatomical MRI will be done for source location. Brain resting state activity will be recorded with MEG/EEG and fMRI.

ELIGIBILITY:
Inclusion Criteria:

* ALS, MRC score ≥ 4 at least in one hand
* Controls: no history of neurological disorders, right-handed

Exclusion Criteria:

* contraindication to MRI

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — controls will be gender and age-matched to ALS
Enrollment: 52 (Actual)
Dates: Start 2018-11-26 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Brain activity | 1 hour
  Brain parametric maps

SECONDARY OUTCOMES:
Brain connectivity | 15 min
  diffusion brain MRI (tractography)

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-Francois Pradat, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Veronique Marchand-Pauvert, PhD, Study Director — Institut National de la Santé Et de la Recherche Médicale, France
Locations (1):
- Hopital Pitie-Salpetriere, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sangari S, Giron A, Marrelec G, Pradat PF, Marchand-Pauvert V. Abnormal cortical brain integration of somatosensory afferents in ALS. Clin Neurophysiol. 2018 Apr;129(4):874-884. doi: 10.1016/j.clinph.2017.12.008. Epub 2017 Dec 24. PMID 29317192
- [Result] Benetton C, Preuilh A, Khamaysa M, Chaumon M, Lackmy-Vallee A, Er A, Pelegrini-Issac M, Querin G, Rouaux C, Pradat PF, Marchand-Pauvert V. Encephalography cross-frequency coupling and brain alteration in amyotrophic lateral sclerosis. Brain Commun. 2025 Jun 6;7(3):fcaf192. doi: 10.1093/braincomms/fcaf192. eCollection 2025. PMID 40488178
- See also: This paper reports results — https://hal.science/hal-04497572v1/file/ISBI24_paper_414.pdf